CLINICAL TRIAL: NCT07363447
Title: The Role of Supervision: Effects of Different Telerehabilitation Methods In Patients With Hypertension
Brief Title: Effects of Different Telerehabilitation Methods In Patients With Hypertension (TELE-HT)
Acronym: TELE-HT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Bozok University (Other)
Responsible Party: Principal Investigator, Beyza Karadüz, PhD Student, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-KAEK-189_2024.02.23_01
Record Dates: First submitted 2026-01-03; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Arterial Hypertension; Systemic Hypertension
Keywords: telerehabilitation; cardiac rehabilitation; Aerobic exercise; synchronous; asynchronous
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Allocation and Sequence: Participants are initially randomly assigned to either the Synchronous Telerehabilitation (STR) or Asynchronous Telerehabilitation (ATR) group using a computer-supported simple randomization procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Telerehabilitation (STR) (Active Comparator): 8-week aerobic-based calisthenics (3 sessions/week, 45 min/session) under real-time physiotherapist supervision via videoconferencing.
  Interventions: Behavioral: Synchronous Cardiac Telerehabilitation
- Asynchronous Telerehabilitation (ATR) (Active Comparator): 8-week aerobic-based calisthenics (3 sessions/week, 45 min/session) delivered via pre-recorded videos and exercise diaries.
  Interventions: Behavioral: Asynchronous Cardiac Telerehabilitation

INTERVENTIONS:
Behavioral: Synchronous Cardiac Telerehabilitation — An 8-week aerobic-based calisthenics program consisting of 24 sessions (3 sessions/week, 45 minutes each).
  Exercises are performed in real-time under the live supervision of a physiotherapist via videoconferencing (WhatsApp).
  Intensity is maintained at 70-85% of age-predicted maximum heart rate, monitored in real-time using a wearable smartband.
  Exercises include high knees, knee-to-elbow, side jacks, and other calisthenics.
  Other Names: Home-based Exercise Training; aerobic exercise training
  Arms: Synchronous Telerehabilitation (STR)
Behavioral: Asynchronous Cardiac Telerehabilitation — The same 8-week aerobic-based calisthenics program (24 sessions, 3 sessions/week) as the STR group.
  Exercises are performed independently by participants using pre-recorded video content.
  Participants maintain an exercise diary to record heart rate and blood pressure levels, which are reviewed weekly by a physiotherapist.
  Exercise intensity is adjusted weekly based on data from the participant's wearable smartband.
  Other Names: Home-based Exercise Training; aerobic exercise training
  Arms: Asynchronous Telerehabilitation (ATR)

SUMMARY:
This study aims to compare two different ways of providing exercise therapy to people with high blood pressure (hypertension) through digital technology. Participants are divided into two groups: one group performs exercises at home while being watched and guided by a physiotherapist in real-time through video calls (synchronous). The other group performs the same exercises by watching pre-recorded videos on their own (asynchronous). The study measures how these two methods affect the patients' exercise capacity, daily blood pressure levels, heart functions, and their ability to manage their own health over an 8-week period.

DETAILED DESCRIPTION:
In this randomized, controlled, single-blinded study, 35 hypertensive individuals are assigned to either a synchronous telerehabilitation (STR) or an asynchronous telerehabilitation (ATR) group. Both groups perform an 8-week aerobic-based calisthenics program consisting of 24 sessions (3 sessions per week, 45 minutes each). The STR group exercises under the live supervision of a physiotherapist via videoconferencing. The ATR group uses pre-recorded video content and maintains an exercise diary. During all sessions, heart rate is monitored in real-time using wearable smartbands to maintain a submaximal intensity (70-85% of age-predicted maximum heart rate). Assessments performed at baseline and at the 8th week include ambulatory blood pressure monitoring (ABPM), transthoracic echocardiography (TTE), maximal stress tests, self-care inventories, physical activity and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic hypertension.
* Age between 18 and 65 years.
* Access to the internet.
* Ownership of a mobile device suitable for telerehabilitation participation.

Exclusion Criteria:

* Presence of comorbid cardiovascular and/or pulmonary diseases.
* Unstable metabolic conditions.
* History of cerebrovascular and/or cardiovascular disease events within the past three months.
* Mental disorders that interfere with exercise cooperation.
* Balance or fall-related problems.
* Orthopedic or neurological conditions that compromise the safety of exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | Before and after the training (0 and 8th Week)
  Change in Functional Exercise Capacity (6-Minute Stepper Test); The number of steps completed within six minutes using a stepper device. Higher step counts indicate better functional capacity.
Exercise Capacity | Before and after the training (0 and 8th weeks)
  Predicted maximal oxygen uptake; Calculated from the duration of the maximal stress test (Bruce protocol) using validated formulas for men and women. It represents maximal aerobic capacity in mL/kg/min.

SECONDARY OUTCOMES:
Blood Pressure Levels | Before and after the training (0 and 8th weeks)
  Ambulatory Blood Pressure Monitoring (ABPM) Parameters; Mean 24-hour, daytime, and nighttime systolic (SBP) and diastolic blood pressure (DBP) levels measured in mmHg.
Cardiac Functions | Before and after the training (0 and 8th weeks)
  Systolic functions assessed with echocardiography expressed by ejection fraction (EF, %) and diastolic functions E and A waves measured via transthoracic echocardiography (TTE). E wave represents early diastolic velocity, and A wave represents late diastolic velocity.
Self-Care Levels | Before and after the training (0 and 8th weeks)
  Self-Care of Hypertension Inventory (SC-HI V3.0) Score; A 23-item Likert-type scale with maintenance, monitoring, and management subscales. Each subscale is scored from 0 to 100, where higher scores indicate better self-care.
Postural Stability and Upper Extremity Function | Before and after the training (0 and 8th weeks)
  Plank test duration (in seconds)
Lower Extremity Muscle Function | Before and after the trainining (0 and 8th weeks)
  Numbers of Squat
Objective Physical Activity Level | Before and after the training (0 and 8th weeks)
  Average daily and weekly total step counts and weekly exercise duration were recorded using a wearable smart wristband
Subjective Physical Activity Levels | Before and after the training (0 and 8th weeks)
  Self-reported PA levels according to the International Physical Activity Questionnaire (IPAQ) score. IPAQ includes vigorous, moderate and walking activities during the last seven days and higher scores reflect higher physical activity levels.
Body Mass Index | Before and after the training (0 and 8th weeks)
  Body weight/ (height*height) (kg/m2)
Body Composition-Anthropometric Measure | Before and after the training (0 and 8th weeks)
  Weight to height ratio (kg/cm)
Body Fat Percantage | Before and after the training (0 and 8th weeks)
  body fat percentage (%) assessed by bioelectrical impedance analysis
Fat Free Mass | Before and after the training (0 and 8th weeks)
  Fat Free Mass assessed by bioelectrical impedance analysis
Lipid Profile | Before and after the training (0 and 8th weeks)
  Measured via blood samples including low-density lipoprotein (LDL) and high-density lipoprotein (HDL) levels in mg/dL.
Cardiovascular Disease (CVD) Risk Profile | Before and after the training (0 and 8the weeks)
  Cardiovascular Disease (CVD) Risk Profile; Estimated using the SCORE-TR risk chart, which calculates the 10-year risk of fatal cardiovascular disease based on age, gender, smoking status, systolic blood pressure, and total cholesterol.
Waist Circumference | Before and after the training (0 and 8th weeks)
  Waist Circumference in cm

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared due to ethical restrictions, institutional policies, and national legal regulations (such as KVKK) regarding the protection of sensitive personal health data in Turkey. The informed consent obtained from participants does not include permission for the public sharing of their raw clinical and diagnostic data.

REFERENCES:
- [Result] Brouwers RWM, Scherrenberg M, Kemps HMC, Dendale P, Snoek JA. Cardiac telerehabilitation: current status and future perspectives. Neth Heart J. 2024 Jan;32(1):31-37. doi: 10.1007/s12471-023-01833-9. Epub 2023 Dec 12. PMID 38085505